CLINICAL TRIAL: NCT00906269
Title: Post-Prostatectomy Erectile Dysfunction: Effect of Hyperbaric Oxygen Therapy
Brief Title: Can Hyperbaric Oxygen Improve Erectile Function Following Surgery for Prostate Cancer
Acronym: HBOT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STAF001982HU
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Impotence; Prostatic Neoplasms
Keywords: impotence; prostatic neoplasms; hyperbaric oxygenation; Phosphodiesterase Inhibitors
MeSH Terms: conditions — Erectile Dysfunction; Prostatic Neoplasms | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Sildenafil therapy plus post-NSRRP HBO2T
- 2 (Sham Comparator)
  Interventions: Drug: Sildenafil therapy plus sham post-NSRRP HBO2T

INTERVENTIONS:
Drug: Sildenafil therapy plus post-NSRRP HBO2T — Sildenafil (Viagra) 50 mg - PO QHS for 12 months beginning the first evening they return home from surgical hospital stay PLUS Post-NSRRP hyperbaric oxygen therapy (90 minutes of 100% oxygen at 2.2ATA (equivalent to the pressure exerted at a depth of approximately 40 feet below sea level). There will be 5 or 10 treatments. The full treatment cycle will be completed within 2 weeks.
  Other Names: Viagra
  Arms: 1
Drug: Sildenafil therapy plus sham post-NSRRP HBO2T — Sildenafil (Viagra)50 mg - PO QHS for 12 months beginning the first evening they return home from surgical hospital stay PLUS Post-NSRRP sham hyperbaric oxygen therapy - 90 minutes at 2.2ATA but instead of 100% oxygen, they will receive air administered via the oxygen hoods, as if they were being administered oxygen. Participants in this group will receive 5 or 10 sham treatment sessions. Full treatment cycle will be completed within 2 weeks.
  Other Names: Viagra
  Arms: 2

SUMMARY:
The purpose of this study is to determine if adding hyperbaric oxygen therapy, a therapy that delivers oxygen under slight pressure, to a drug treatment of PDE5I (such as Viagra, Levitra, Cialis)for men following surgery for prostate cancer will result in more men being able to continue to have erections.

DETAILED DESCRIPTION:
Prostate cancer is the most common non-skin malignancy in men in the United States, with approximately 232,000 diagnoses of adenocarcinoma projected for 2005. More than 150,000 of these men are treated with radical prostatectomy. Common sequelae following successful NSRRP (nerve-sparing radical retropubic prostatectomy)include urinary incontinence and sexual dysfunction. Recent advances in surgery technique and treatment have been made but in spite of aggressive management, recovery of sexual function is incomplete with fewer than one-fifth reporting return to baseline. The etiology of erectile dysfunction following radical prostatectomy results most probably from local surgical trauma and neurapraxia, which leads to corpus cavernosal hypoxemia in the post-NSRRP period. This hypoxemia is believed to impact negatively on the health and maintenance of the smooth muscle cells within the corpus cavernosum. Hyperbaric oxygen therapy (HBO2T) is a unique modality that is able to provide oxygen delivery to tissues that have been damaged by traumatic injury.

Hypothesis: The addition of post-NSRRP hyperbaric oxygen therapy (HBO2T) to a treatment of phosphodiesterase type 5 inhibitor (PDE5I) will reduce the incidence of erectile dysfunction (ED) and urinary incontinence when measured at 1, 3, 6, 12 and 18 months post-NSRRP for Stage I prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* male
* age 40-69
* diagnosis of Stage I prostate cancer
* bilateral NSRRP as primary treatment
* sexual potency prior to surgery

Exclusion Criteria:

* COPD, CHF, diabetes mellitus
* known inability to tolerate PDE5I
* confinement anxiety/claustrophobia
* planned adjuvant or neo-adjuvant therapy
* patients taking alpha blockers or nitrates
* patients with retinitis pigmentosa

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-07; Primary Completion 2020-07 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Erectile function domain of Internation Index of Erectile Function (IIEF) | 1, 3, 6, 12, and 18 months post surgery

SECONDARY OUTCOMES:
clinical or biochemical recurrence of cancer | up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: James Graydon, MD, Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

REFERENCES:
- [Background] Burnett AL. Erectile dysfunction following radical prostatectomy. JAMA. 2005 Jun 1;293(21):2648-53. doi: 10.1001/jama.293.21.2648. PMID 15928287
- [Background] Mulhall JP, Graydon RJ. The hemodynamics of erectile dysfunction following nerve-sparing radical retropubic prostatectomy. Int J Impot Res. 1996 Jun;8(2):91-4. PMID 8858398
- [Background] Walsh PC, Donker PJ. Impotence following radical prostatectomy: insight into etiology and prevention. J Urol. 1982 Sep;128(3):492-7. doi: 10.1016/s0022-5347(17)53012-8. No abstract available. PMID 7120554
- [Background] Rosen RC, Riley A, Wagner G, Osterloh IH, Kirkpatrick J, Mishra A. The international index of erectile function (IIEF): a multidimensional scale for assessment of erectile dysfunction. Urology. 1997 Jun;49(6):822-30. doi: 10.1016/s0090-4295(97)00238-0. PMID 9187685
- [Background] Wei JT, Dunn RL, Litwin MS, Sandler HM, Sanda MG. Development and validation of the expanded prostate cancer index composite (EPIC) for comprehensive assessment of health-related quality of life in men with prostate cancer. Urology. 2000 Dec 20;56(6):899-905. doi: 10.1016/s0090-4295(00)00858-x. PMID 11113727
- [Background] Feldmeier, J.J.,Chairman and Editor. Hyperbaric Oxygen 2003: Indications and Results. The Hyperbaric Oxygen Therapy Committee Report . Kensington, MD: Undersea and Hyperbaric Medicine Society, 2003.
- [Background] Feldmeier JJ. Hyperbaric oxygen: does it have a cancer causing or growth enhancing effect? In: Proceeding of the Concensus Conference sponsored by the European Society for Therapeutic Radiology and Oncology and the European Committee for Hyperbaric Medicine. Portugal 2001: 129-146
- [Result] Link RE, Su LM, Sullivan W, Bhayani SB, Pavlovich CP. Health related quality of life before and after laparoscopic radical prostatectomy. J Urol. 2005 Jan;173(1):175-9; discussion 179. doi: 10.1097/01.ju.0000147190.67218.1b. PMID 15592069
- [Result] Zamboni WA, Brown RE, Roth AC, Mathur A, Stephenson LL. Functional evaluation of peripheral-nerve repair and the effect of hyperbaric oxygen. J Reconstr Microsurg. 1995 Jan;11(1):27-9; discussion 29-30. doi: 10.1055/s-2007-1006507. PMID 7714876
- [Result] Kaufman JM, Graydon RJ. Androgen replacement after curative radical prostatectomy for prostate cancer in hypogonadal men. J Urol. 2004 Sep;172(3):920-2. doi: 10.1097/01.ju.0000136269.10161.32. PMID 15310998
- [Result] Lowentritt BH, Scardino PT, Miles BJ, Orejuela FJ, Schatte EC, Slawin KM, Elliott SP, Kim ED. Sildenafil citrate after radical retropubic prostatectomy. J Urol. 1999 Nov;162(5):1614-7. PMID 10524880
- [Result] Schwartz EJ, Wong P, Graydon RJ. Sildenafil preserves intracorporeal smooth muscle after radical retropubic prostatectomy. J Urol. 2004 Feb;171(2 Pt 1):771-4. doi: 10.1097/01.ju.0000106970.97082.61. PMID 14713808
- See also: Hartford Hospital Home Page — http://www.harthosp.org